CLINICAL TRIAL: NCT01865916
Title: 2L Oral Bi-PegLyte Versus 2L Oral MoviPrep Regimen for Outpatient Colonic Preparation: A Randomized, Non-Inferiority Open Trial
Brief Title: 2L Oral Bi-PegLyte Versus 2L Oral MoviPrep Regimen for Outpatient Colonic Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H13-00502
Record Dates: First submitted 2013-05-13; First posted 2013-05-31 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; Bisacodyl; Ascorbic Acid; MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 Liters Bi-Peglyte (Active Comparator): Subjects will be asked to take split dose of 2 Liters PEG + 15mg bisacodyl for bowel preparation the day before colonoscopy.
  Interventions: Drug: Polyethylene Glycol (PEG) and 15 mg Bisacodyl
- 2 Liters Moviprep (Experimental): Subject will be asked to take split dose of 2 Liters PEG + ascorbic acid for bowel preparation the day before colonoscopy
  Interventions: Drug: Polyethylene Glycol (PEG) + ascorbic acid

INTERVENTIONS:
Drug: Polyethylene Glycol (PEG) and 15 mg Bisacodyl — Subjects will be asked to take split dose of 2L PEG and 3 tablets of 5 mg Bisacodyl
  Other Names: Bi-Peglyte
  Arms: 2 Liters Bi-Peglyte
Drug: Polyethylene Glycol (PEG) + ascorbic acid — Subjects will be asked to take split dose of 2L PEG and vitamin C
  Other Names: Moviprep
  Arms: 2 Liters Moviprep

SUMMARY:
This study is a randomized, controlled, single centre, endoscopist-blinded non-inferiority trial. The purpose of our study is to determine if using a 2-litre mixture in combination with vitamin C is better than using 2 litres of mixture with bisacodyl tablets. Two-litre PegLyte based preparations with an added laxative agent are commonly used for colonoscopies in outpatient settings. If the investigators discover that a 2-litre mixture with either the tablets or the ascorbic acid work better, future patients undergoing colonoscopy will be able to experience fewer side effects and be less troubled by the preparation while still allowing a good view of the colon.

DETAILED DESCRIPTION:
All adults (≥ 19 yrs of age) who are referred to St. Paul's Hospital for outpatient colonoscopy will be included in our study. Exclusion criteria included those with constipation, suspected or known small bowel obstruction, severe inflammatory bowel disease, and any history of colonic resection. 278 consecutive eligible patients will be randomized to one of two bowel preparations through the use of concealed allocation by a scheduling assistant (blinded) in a one-to-one allocation ratio. Bowel preparations included: (i) 2 L of MoviPrep (2 L PEG 3350 electrolyte solution + ascorbic acid) or (ii) Bi-Peglyte (2 L PEG 3350 electrolyte solution and 15mg bisacodyl). Patients in both arms will be instructed to adhere to a clear liquid diet commensing 24 hours prior to scheduled colonoscopy in addition to their remaining bowel preparation.

The investigators will not have access to the randomization envelopes and the randomized bowel preparation will be stored within the medical record that will not be accessible by the endoscopist. The endoscopists can break blinding and access the bowel prep given when medically necessary.

At the time of their procedure check-in, written consent will be confirmed and patients will respond to a brief survey assessing patient tolerance. All colonoscopies will be performed under conscious sedation by an experienced endoscopist. Endoscopists will be blinded to the bowel preparation until the completion of the study. We will use the Boston Bowel Preparation Scale (BBPS) and Ottawa Bowel Preparation Scale (OBPS) to assess efficacy in bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* All adults (≥ 19 years of age) who are referred to St. Paul's Hospital for outpatient colonoscopy will be included in our study.

Exclusion Criteria:

* those with constipation,
* suspected or known small bowel obstruction,
* severe inflammatory bowel disease, and
* any history of colonic resection.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing efficacy as rated by a Boston Bowel Preparation Scale score of greater than 8 | 20 hours
  The BBPS is a relatively new, validated scoring system assessing cleanliness of three segments of the colon (left colon, transverse, and right colon). The total is a 10 point scale (0-9) that grades each segment of the colon from 0-3. A segment score of 0 describes: 'unprepared colon segment with mucosa not well seen due to solid stool that cannot be cleared'. Segment score 1: 'portion of mucosa of the colon segment seen, but other areas of the colon are not well seen due to staining, residual stool and/or opaque liquid'. Segment score 2: 'minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well'. Segment score 3: 'entire mucosa of the colon segment seen well with no residual staining, small fragments of stool and/or opaque liquid'. In this study, we define an excellent equivalent BBPS score as 8 or 9. Scores of 7 or above are generally felt to provide a good visualization of the colon.

SECONDARY OUTCOMES:
Patient tolerability to each 2L product | 20 hours
  Our secondary outcome is patient tolerability to each 2L product based on a ten-question survey. The questionnaire basically asks about patient experience in terms of charateristic taste of bowel prep, volume intake, any distressing signs and symptoms, compliance to bowel preparation solution assigned to subjects using a Likert scale. The number of participants in each level will subsequently be quantified (n,%) and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, MD, FRCP, Principal Investigator — University of British Columbia
Locations (1):
- GI Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Beck DE, Harford FJ, DiPalma JA. Comparison of cleansing methods in preparation for colonic surgery. Dis Colon Rectum. 1985 Jul;28(7):491-5. doi: 10.1007/BF02554091. PMID 4017808
- [Background] American Society of Colon and Rectal Surgeons (ASCRS); American Society for Gastrointestinal Endoscopy (ASGE); Society of American Gastrointestinal and Endoscopic Surgeons (SAGES); Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE. A consensus document on bowel preparation before colonoscopy: prepared by a task force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Surg Endosc. 2006 Jul;20(7):1147-60. doi: 10.1007/s00464-006-0152-y. Epub 2006 Jun 8. No abstract available. PMID 16763922
- [Background] Hsu CW, Imperiale TF. Meta-analysis and cost comparison of polyethylene glycol lavage versus sodium phosphate for colonoscopy preparation. Gastrointest Endosc. 1998 Sep;48(3):276-82. doi: 10.1016/s0016-5107(98)70191-9. PMID 9744604
- [Background] Curran MP, Plosker GL. Oral sodium phosphate solution: a review of its use as a colorectal cleanser. Drugs. 2004;64(15):1697-714. doi: 10.2165/00003495-200464150-00009. PMID 15257632
- [Background] Vanner SJ, MacDonald PH, Paterson WG, Prentice RS, Da Costa LR, Beck IT. A randomized prospective trial comparing oral sodium phosphate with standard polyethylene glycol-based lavage solution (Golytely) in the preparation of patients for colonoscopy. Am J Gastroenterol. 1990 Apr;85(4):422-7. PMID 2183591
- [Background] Frommer D. Cleansing ability and tolerance of three bowel preparations for colonoscopy. Dis Colon Rectum. 1997 Jan;40(1):100-4. doi: 10.1007/BF02055690. PMID 9102248
- [Background] Davis GR, Santa Ana CA, Morawski SG, Fordtran JS. Development of a lavage solution associated with minimal water and electrolyte absorption or secretion. Gastroenterology. 1980 May;78(5 Pt 1):991-5. PMID 7380204